CLINICAL TRIAL: NCT04529018
Title: A Phase 1 Clinical Trial Evaluating the Safety and Efficacy of up to Two Administrations of the Adrenal PET Tracer [18F]CETO in Healthy Volunteers and Patients With Primary Aldosteronism
Brief Title: CETO First in Human Trial
Acronym: CETO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Professor Mark Gurnell, Professor in Clinical Endocrinology and Honorary Consultant, University of Cambridge
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CETO-FIH; 2018-004851-18 (EudraCT Number); ISRCTN16159564 (Other: ISRCTN registry)
Record Dates: First submitted 2020-08-13; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Primary Aldosteronism
Keywords: Adrenal; Conn's; Endocrine; Aldosterone
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Intervention Model Description: Phase I single-centre, open-label, micro-dosing study
Who Masked: Outcomes Assessor
Masking Description: Scans will be assessed by two independent nuclear medicine physicians, who will be blinded to patient identifiable data when analysing PET-CT scans.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (Experimental): A group of 5 healthy volunteers will be tested with the PET radiotracer [18F]CETO to assess safety of tracer administration, and evaluate uptake by the normal adrenal glands.
  Interventions: Combination Product: [18F]CETO
- Patients with primary aldosteronism (Experimental): A group of 6 patients with Primary Aldosteronism (3 with unilateral and 3 with bilateral disease) will be tested with up to two administrations of the PET radiotracer [18F]CETO, to assess safety of tracer administration, evaluate the ability of [18F]CETO to distinguish between unilateral and bilateral cases of PA, and determine the effect of Dexamethasone in improving the quality of PET-CT images acquired following administration.
  Interventions: Combination Product: [18F]CETO

INTERVENTIONS:
Combination Product: [18F]CETO — [18F]CETO is a PET radiotracer used to diagnose and visualise the cause(s) of primary aldosteronism
  Other Names: CETO

SUMMARY:
The study is a Phase 1, single-centre, open label, micro-dosing study. The aim is to investigate an innovative new tracer, [18F]CETO, as a potential alternative to adrenal vein sampling for the lateralisation of primary aldosteronism (PA).

DETAILED DESCRIPTION:
At least one-quarter of the UK adult population has hypertension, a major risk factor for heart attacks and stroke. Primary aldosteronism (PA), a treatable form of hypertension, accounts for 5-10% of all cases, and 20-25% of difficult to control hypertension. It is challenging to determine whether one adrenal gland is the source of PA (which is potentially curable with surgery) or both glands (which would require long-term drug treatment). Existing lateralising procedures (i.e. investigations to distinguish one from two gland involvement e.g. CT or MRI scan) have significant limitations. Accordingly, most patients must undergo an invasive procedure called adrenal vein sampling (AVS) in which small catheters are placed in each adrenal vein. However, this is time-consuming, technically demanding, and fails in 20-50% of cases. To address this, researchers have adopted a novel approach using PET-CT as an alternative to AVS. Currently, this uses a tracer called metomidate labelled with carbon-11 (11C MTO), which is taken up preferentially by the adrenal gland, and in particular by adrenal tumours causing PA. However, its utility is limited by a short half-life, which means the scan can only be performed in centres with a cyclotron facility (currently less than 10 NHS sites). The aim of this study is to investigate the safety of a new tracer with a longer half-life, [18F]CETO, that could be made available for use in many more centres.

The trial objectives are outlined below:

Primary Objective

To evaluate the safety of up to two administrations of [18F]CETO in up to 6 patients with primary aldosteronism and 5 healthy volunteers.

Secondary Objective

* Assess [18F]CETO uptake by the adrenal glands
* Evaluate uptake in bilateral vs unilateral cases of PA following [18F]CETO administration in up to 6 patients.

ELIGIBILITY:
Healthy Volunteers

To be included in the trial the participant must:

* give written informed consent
* be aged 50 years or over
* have no underlying medical conditions
* be able to lie down for at least 2 hours and not be claustrophobic

In addition, all female participants must be:

- post-menopausal (no menses for 12 months, without an alternative medical cause)

Patients

To be included in the trial the patient must:

* give written informed consent
* be aged 40 years or over
* be able to lie down for at least 2 hours and not be claustrophobic

fulfil the following criteria:

* have a confirmed diagnosis of PA as per Endocrine Society guidelines
* At least one paired measurement of plasma renin and aldosterone, measured off Spironolactone/Eplerenone within past 12 months, showing ARR above local threshold value.
* One of the following two criteria:
* Plasma aldosterone>190pmol/L following saline infusion.
* Spontaneous hypokalaemia, suppressed plasma renin and plasma aldosterone>550pmol/L.
* have undergone successful lateralisation of the cause of PA to one or both adrenal glands by adrenal vein sampling (AVS).
* be willing to have two scans

In addition, all female patients must have a negative (blood) pregnancy test at the screening visit.

Exclusion Criteria:

All participants:

* allergy to radiographic contrast agents
* allergy or contraindication to synacthen
* pregnancy, breastfeeding, or the intention to become pregnant during the 6 months following trial participation
* positive pregnancy test at the screening or baseline visits
* assessed by the investigator as being unable or unwilling to comply with the requirements of the study protocol.
* receipt of another IMP as part of a CTIMP
* prior radiation exposure as part of previous research studies
* recreational drug use, or substance/alcohol dependency
* clinically abnormal screening blood tests.

Additional exclusion criteria for healthy volunteers:

* women of child-bearing potential (i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile)
* exposure to radiation during their work
* received more than 10 mSv of radioactivity in the past 12 months
* any subject with a history of adrenal disease or who, at the screening visit, reports symptoms, or exhibits physical signs, that could be consistent with previously unsuspected adrenal disease

Additional exclusion criteria for patients:

- allergy or contraindication to dexamethasone treatment (or lactose intolerant)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety of [18F]CETO administration | 6 months
  The primary outcome measure is the overall safety of [18F]CETO. This will be assessed according to the frequency of adverse events, serious adverse events, clinically significant changes in vital signs, ECG and laboratory parameters.

SECONDARY OUTCOMES:
[18F]CETO uptake by the the adrenal glands. | 6 months
  [18F]CETO uptake by the adrenal glands will be assessed by measurement of Standardized Uptake Values (SUV) over the left and right adrenal glands. All assessments will be performed by a dedicated blinded reviewer.
To evaluate uptake in bilateral versus unilateral cases of PA following [18F]CETO administration in up to 6 patients. | 6 months
  Evaluation of adrenal uptake of [18F]CETO in bilateral versus unilateral cases of PA will be performed by comparing SUV values of both adrenal glands in three patients with each subtype of PA (using a dedicated blinded reviewer).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gurnell, PhD, FRCP, Principal Investigator — University of Cambridge
Locations (1):
- Addenbrooke' Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burton TJ, Mackenzie IS, Balan K, Koo B, Bird N, Soloviev DV, Azizan EA, Aigbirhio F, Gurnell M, Brown MJ. Evaluation of the sensitivity and specificity of (11)C-metomidate positron emission tomography (PET)-CT for lateralizing aldosterone secretion by Conn's adenomas. J Clin Endocrinol Metab. 2012 Jan;97(1):100-9. doi: 10.1210/jc.2011-1537. Epub 2011 Nov 23. PMID 22112805
- [Background] Hahner S, Stuermer A, Kreissl M, Reiners C, Fassnacht M, Haenscheid H, Beuschlein F, Zink M, Lang K, Allolio B, Schirbel A. [123 I]Iodometomidate for molecular imaging of adrenocortical cytochrome P450 family 11B enzymes. J Clin Endocrinol Metab. 2008 Jun;93(6):2358-65. doi: 10.1210/jc.2008-0050. Epub 2008 Apr 8. PMID 18397978
- [Background] Bergstrom M, Juhlin C, Bonasera TA, Sundin A, Rastad J, Akerstrom G, Langstrom B. PET imaging of adrenal cortical tumors with the 11beta-hydroxylase tracer 11C-metomidate. J Nucl Med. 2000 Feb;41(2):275-82. PMID 10688111